CLINICAL TRIAL: NCT01497457
Title: Interest of Saline MR Peritoneography for Pre-operative Assessment of Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B403201112604
Record Dates: First submitted 2011-12-14; First posted 2011-12-22 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR saline peritoneography (Experimental): Patients that will undergo MR saline peritoneography
  Interventions: Procedure: MR saline peritoneography

INTERVENTIONS:
Procedure: MR saline peritoneography — Ultrasound-guided Intraperitoneal injection of 250cc of steril saline solution with a 22G needle, followed by rectal MR imaging

SUMMARY:
MR saline peritoneography could be useful to demonstrate the peritoneal outline of the pouch of Douglas. The investigators think that the localization of the rectal tumor in function of this anatomic mark could be decisive for pre-operative assessment.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma

Exclusion Criteria:

* Metastatic disease
* under 18y patient
* woman of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determination of the distance between a rectal tumor and the pouch of Douglas | Two years
  Feasability of the determination of the distance between a rectal tumor and the pouch of Douglas by MR saline peritoneography:
  1. Visualisation of the Douglas
  2. Visualisation of the Tumor
  3. Determination of the distance between the tumor and the pouch of Douglas

CONTACTS AND LOCATIONS:
Overall Officials: Cristina A Dragean, MD, Principal Investigator — Cliniques Universitaires St Luc - Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires St Luc - Université Catholique de Louvain, Brussels, Belgium